CLINICAL TRIAL: NCT02558608
Title: Effect of Dissecting of The Inferior Pulmonary Ligament on Postoperative Pulmonary Reexpansion and Recurrence After Operation by Video-assisted Thoracic Surgery in the Treatment of Primary Spontaneous Pneumothorax(PSP)
Brief Title: Effect of Dissecting of The Inferior Pulmonary Ligament on Postoperative Pulmonary Reexpansion and Recurrence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Principal Investigator, Jian Cui, Principal Investigator, Beijing Haidian Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPL001
Record Dates: First submitted 2015-09-13; First posted 2015-09-24 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Pneumothorax
Keywords: Prime Spontaneous Pneumothorax; recurrence
MeSH Terms: conditions — Pneumothorax; Recurrence | interventions — Thoracoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WR AND DIPL (Experimental): patients undergo wedge resection and dissection the inferior pulmonary ligament by thoracoscopic surgery or video assisted thoracoscopic surgery
  Interventions: Procedure: DIPL; Procedure: WR; Procedure: thoracoscopic surgery
- WR (Active Comparator): patients undergo wedge resection by thoracoscopic surgery or video assisted thoracoscopic surgery without dissection the inferior pulmonary ligament
  Interventions: Procedure: WR; Procedure: thoracoscopic surgery

INTERVENTIONS:
Procedure: DIPL — dissection of the inferior pulmonary ligament
  Arms: WR AND DIPL
Procedure: WR — wedge resection of the lung bleb
Procedure: thoracoscopic surgery — surgery performed by video assisted thoracoscopy

SUMMARY:
This subject analysis of the influence of the dissociating inferior pulmonary ligament on pulmonary reexpansion and recurrence in the treatment of primary spontaneous pneumothorax by video assisted thoracic surgery. All patients are randomly divided into two groups: group A and group B. Wedge resection(WR) will be performed for all patients. Investigators dissect the inferior pulmonary ligament(DIPL) for group A. Investigators do not dissect the inferior pulmonary ligament for group B. The pulmonary reexpansion and recurrence rate are observed between the two groups.

DETAILED DESCRIPTION:
Wedge resection of the lung is usually used in the treatment of primary spontaneous pneumothorax. And the pleural treatment also might be used. But part of secondary pneumothorax patients who had undergone surgical, the bullae can be found especially in the apical of lung, even if the pleural have been treated in some way.This subject provides a new way of thinking and method to solve the problem of recurrent spontaneous pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

1. The patients diagnosis pneumothorax with chest radiograph or computed tomography (CT)
2. The clinical and final pathological diagnosis for patient is PSP.
3. The patients with stable vital signs, no contraindication for operation and no communication barriers.
4. The patients,after informed of test content, significance and risk, who voluntarily enroll and sign informed consent.

Exclusion Criteria:

1. The patients who refuse to do a video assisted thoracic surgery.
2. The patients with pneumothorax with specific causes such as pulmonary hamartoangiomyomatosis, catamenial pneumothorax, and pneumothorax secondary to chronic obstructive pulmonary disease.
3. The patients who were older than 50 years
4. The patients with familial history of pneumothorax.
5. The patients with mental disorders, low Intelligence Quotient, can not objectively reflect the indicators of observation.
6. The patients who refuse to follow-up.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | 3 years
  the 3- year recurrence rate of pneumothorax after surgery.

SECONDARY OUTCOMES:
pulmonary reexpansion rate | 1 day and 4 days
  the proportion of pulmonary reexpansion on the first and fourth day after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Cui, director, Study Director — Beijing Haidian Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest. 2001 Feb;119(2):590-602. doi: 10.1378/chest.119.2.590. PMID 11171742
- [Background] Gaunt A, Martin-Ucar AE, Beggs L, Beggs D, Black EA, Duffy JP. Residual apical space following surgery for pneumothorax increases the risk of recurrence. Eur J Cardiothorac Surg. 2008 Jul;34(1):169-73. doi: 10.1016/j.ejcts.2008.03.049. Epub 2008 May 1. PMID 18455414
- [Background] Casali C, Stefani A, Ligabue G, Natali P, Aramini B, Torricelli P, Morandi U. Role of blebs and bullae detected by high-resolution computed tomography and recurrent spontaneous pneumothorax. Ann Thorac Surg. 2013 Jan;95(1):249-55. doi: 10.1016/j.athoracsur.2012.05.073. Epub 2012 Jul 10. PMID 22785214
- [Background] Min X, Huang Y, Yang Y, Chen Y, Cui J, Wang C, Huang Y, Liu J, Wang J. Mechanical pleurodesis does not reduce recurrence of spontaneous pneumothorax: a randomized trial. Ann Thorac Surg. 2014 Nov;98(5):1790-6; discussion 1796. doi: 10.1016/j.athoracsur.2014.06.034. Epub 2014 Sep 16. PMID 25236367
- [Background] Hatz RA, Kaps MF, Meimarakis G, Loehe F, Muller C, Furst H. Long-term results after video-assisted thoracoscopic surgery for first-time and recurrent spontaneous pneumothorax. Ann Thorac Surg. 2000 Jul;70(1):253-7. doi: 10.1016/s0003-4975(00)01411-9. PMID 10921718